CLINICAL TRIAL: NCT00654394
Title: Randomized, Double-Blind, Multicenter, Trial to Assess the Effect of High & Low Doses of ZD4522 on Progression of Carotid Artery Atheroma in Moderately Hypercholesterolemic Subjects With Asymptomatic Carotid Stenosis After 24 Months of Dosing.
Brief Title: Progression of Carotid Artery Atheroma in Moderately Hypercholesterolemic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4522IL/0044; D3560C00044
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Carotid Artery Stenosis; Hypercholesterolemia
Keywords: Cholesterol; Carotid Artery Stenosis; Hypercholesterolemia; Rosuvastatin; Crestor
MeSH Terms: conditions — Carotid Stenosis; Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor

SUMMARY:
The purpose of this study is to examine the changes in the carotid artery when subjects receive high or low doses of rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood low density lipoprotein cholesterol level as defined by the protocol
* Diagnosed carotid arterial stenosis

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Heavy or total occlusion of the carotid artery or recent stroke
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2000-01; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Changes in carotid wall volume as measured by MRI scan | At 40 weeks and 104 weeks

SECONDARY OUTCOMES:
Safety: adverse events & abnormal laboratory markers | 2 weekly for first 4 weeks then 4 weekly
Other changes in the structure and composition of the carotid arterial wall as defined in the protocol. | At 40 weeks and 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hatsukami, Principal Investigator — University of Washington, USA; Russell Esterline, Study Director — AstraZeneca

REFERENCES:
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307